CLINICAL TRIAL: NCT04527783
Title: The Use of an Engineered Glove for the Assessment and Rehabilitation of Manual Dexterity in People With Stroke: a Pilot Randomized Control Trial.
Brief Title: The Use of an Engineered Glove for the Assessment and Rehabilitation of Manual Dexterity in People With Stroke.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Davide Cattaneo, Principal Investigator, Fondazione Don Carlo Gnocchi Onlus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GREVAP
Record Dates: First submitted 2020-08-19; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Stroke; Hand Grasp
MeSH Terms: conditions — Stroke | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Each subject will perform a variety of VR exercises to reduce impairments in their finger range of motion, speed and strength.
  It includes a glove-shaped sensor device and a software application.
  Interventions: Other: experimental group
- control group (Active Comparator): Each subject will perform usual care rehabilitation aimed at improving manual dexterity
  Interventions: Other: control group

INTERVENTIONS:
Other: experimental group — Each subject will undergo 10 rehabilitation sessions 2-3 times a week, lasting around 30'.
  Arms: experimental group
Other: control group — Each subject will undergo 10 rehabilitation sessions 2-3 times a week, lasting around 30'.
  Arms: control group

SUMMARY:
Stroke often results in impairments of upper extremity, including coordination deficits, reducing of force, weakness and changes in the kinetic and kinematic workspace of fingers with 75% of stroke survivors facing difficulties performing activities of daily living.

The ability to oppose the fingertip of the thumb to each fingertip of the same hand is the basis of grasping objects of various sizes and operating tools and assessing and improving distal upper extremity function is of primary goal in the rehabilitation of stroke survivors. Moreover, repetitive movement practice seems to be crucial for maximizing therapeutic benefits.

Recent studies, proposed an engineered glove to assess motor performance during finger-to-thumb opposition movements and to provide objective and reproducible measures.

The same tool can be integrated with Virtual Reality and serious games to provide repetitive practice of activities improving motivation and adherence with therapy.

the investigators developed a new integrated glove and virtual reality to facilitate the recovery of hand functionality.

The aim of this study is to investigate the feasibility of the engineered glove in the assessment and treatment of hand dysfunction in people with Stroke.

ELIGIBILITY:
Inclusion Criteria:

* a single stroke,
* some movement of the fingers,
* any technical and difficulties with wearing the glove on the paretic hand

Exclusion Criteria:

* visual or cognitive deficits that would prevent them for performing the task

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Box and Blocks Test | baseline- immediately after the intervention
  Block and Box Test assesses grasp and transport and upper limb functional disorders and measures unilateral gross manual dexterity.

SECONDARY OUTCOMES:
Change in 9-Hole Peg Test | baseline- immediately after the intervention
  It measures finger dexterity. Patient takes the pegs from a container and place them into the holes as quickly as possible.
Change in Manual Ability Measurement | baseline- immediately after the intervention
  It is a self reported questionnaire to rate perceived manual ability on a scale ranging from 0 (impossible to complete any of activity cited) to 100 (every activity cited is accomplished without any difficulty).
Change in the instrumented indexes | baseline- immediately after the intervention
  Subjects perform a repetitive finger-to-thumb opposition sequence (index, medium, ring and little finger) with their affected hand at maximal velocity and with the two hands simultaneously at a frequency of 2 Hz paced by a metronome. The testing session includes one 60sec trial per condition.
  They wear a sensor-engineered glove on both hands to quantitatively assess finger motor performance

IPD SHARING:
Plan to Share IPD: No